CLINICAL TRIAL: NCT07195006
Title: Early Life Diarrhoea Episode(s), Malnutrition, Environmental Enteric Dysfunction and Microbiome Trajectories From Birth Until 3 Years of Life ; The University of Zimbabwe Birth Cohort Study-2 (UZBCS-2)
Brief Title: Early Life Malnutrition, Environmental Enteric Dysfunction and Microbiome Trajectories
Acronym: UZBCS-2
Status: Recruiting | Type: Observational
Sponsor: University of Zimbabwe (Other)
Collaborators: University of Bern (Other); Insel Gruppe AG, University Hospital Bern (Other); LMU Klinikum (Other)
Responsible Party: Sponsor
Other Study IDs: MRCZ/A/3256; JREC/451/2024 (Other: JREC Institutional Ethical Committee)
Record Dates: First submitted 2025-07-18; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Malnutrition Pregnancy; Malnutrition in Children; Malnutrition (Calorie); Environmental Enteric Dysfunction; Gut Dysbiosis; Gut Permeability, Gut Inflammation; Diarrhea Infectious; Maternal Stress; Child Mental Health; Natural Killer Cell Mediated Immunity; Mycotoxin Biomonitoring; Environmental Exposures; Cell-Mediated Immune Deficiency
Keywords: diarrhoeal episodes; short chain fatty acids receptor agonists; intestinal inflammation, leakage and calory extraction; toxins in drinking water and food; macro- and micronutrient composition of breast milk; human anti-Gal antibodies; mitochondria health and nutrient uptake; endothelial dysfunction and oxidative stress; hormonal mediated molecular signalling mechanisms; interaction of epigenetics & socioeconomic factors; microbiota, pathobionts and oral microbiota; metagenomics; undernutrition and intestinal infections; infant mortality, morbidity within 1st 1000 days of life; low mid upper arm circumference; sleep adequacy in maternal mental health; chronic inflammation
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition; Dysentery; Infant Death | interventions — Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Breast milk Stool Mid stream urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group 1; Malnourished pregnant women, improved WASH living conditions: Malnourished, improved WASH: Pregnant women (≥20 weeks) with MUAC ≤23 cm, residing in improved WASH area (Kuwadzana research site, Harare)
  Interventions: Other: Malnutrition in pregnancy as exposure
- Group 2; Normo-nourished pregnant women, improved WASH living conditions: Normo-nourished women, improved WASH living conditions: Pregnant women (≥20 weeks) with MUAC 25-35 cm and Hb ≥11 g/dL, residing in improved WASH area (Kuwadzana research site, Harare)
- Group 3; Malnourished pregnant women, poor WASH living conditions: Malnourished women, poor WASH: Pregnant women (≥20 weeks) with MUAC ≤23 cm, residing in poor WASH area (Hopley research site, Harare)
  Interventions: Other: Malnutrition in pregnancy as exposure; Other: Poor WASH living conditions as exposure
- Group 4; Normo-nourished pregnant women, poor WASH living conditions: Normo-nourished women, poor WASH: Pregnant women (≥20 weeks) with MUAC 25-35 cm and Hb ≥11 g/dL, residing in poor WASH area (Hopley research site, Harare)
  Interventions: Other: Poor WASH living conditions as exposure

INTERVENTIONS:
Other: Malnutrition in pregnancy as exposure — MUAC ≤23 cm in pregnancy at least 20 weeks gestational age
  Groups: Group 1; Malnourished pregnant women, improved WASH living conditions; Group 3; Malnourished pregnant women, poor WASH living conditions
Other: Poor WASH living conditions as exposure — Poor water (source, quality, access, reliability), sanitation (toilet type, cleanliness, number of people using toilet) and personal (hand wash practices) and household hygiene (dumpster availability and emptying frequency) index scores.
  WASH Index score ranges; 1.Basic services (76-100%), 2.Semi-basic services (51-75%) 3.Poor services (26-50%) 4.No services (0-25%)
  Groups: Group 3; Malnourished pregnant women, poor WASH living conditions; Group 4; Normo-nourished pregnant women, poor WASH living conditions

SUMMARY:
Malnutrition in women of reproductive age remains a public health concern in Sub-Saharan Africa (SSA). Malnutrition during pregnancy affects foetal growth with a tendency of the exposed infants to also develop it. The interaction of the mother with the infant shapes the seeding and the trajectory of the infant intestinal microbiota which is crucial for development of a healthy immune system Malnutrition has been associated with intestinal inflammation, intestinal leakage and reduced calorie absorption. Early life malnutrition and environmental enteric dysfunction (EED) immunopathology remains poorly described in the context of mother-infant dyads. This is essential as malnutrition, poor water, sanitation and hygiene (WASH), including the presence of infectious diseases limit the developmental potential of the exposed infants in SSA, including Zimbabwe. In addition, maternal stress and poor mental health may also affect standard hygiene practices, including how a mother cares for her baby, potentially aggravating EED and the risk of the infant being malnourished.

Primary outcomes

1. Infant malnutrition and recovery.
2. Gut dysfunction (gut inflammation, leaky gut, malabsorption, dysbiosis)
3. Diarrhea episodes, defined as any episode of acute diarrhoea (≥3 passages of loose stool within 24 hours as reported by the mother) occurring before the next study visit.

Definition of malnutrition outcomes to be assessed in babies born to malnourished women, is a mid- upper arm circumference (MUAC) <23cm;

* MUAC for age: Malnourished defined as those below -2 standard (SD) of the World Health Organisation (WHO) reference
* Weight-for-age: Underweight defined as those below -2SD WHO reference
* Weight-for-height: Wasted defined as those below -2SD WHO reference
* Height-for-age: Stunted defined as those below -2SD WHO reference
* Z-scores (as they are i.e. a continuous variable, taking age of infants into account)
* A composite variable, any of malnourished, underweight, wasted or stunted.

DETAILED DESCRIPTION:
Background Malnutrition, poor hygiene, lack of access to clean water, infectious diseases, and low access to medicine limit life expectancy and developmental potential of infants in Sub-Saharan Africa (SSA) including Zimbabwe. These conditions severely affect infant growth and neurodevelopment, especially within the first 1000 days of life, and the affected infants might never reach their full development potential in life. The interaction of the mother with the infant shapes the trajectory of the intestinal microbiota and the development of its immune system is considered crucial for a healthy development, yet the therapeutic success remains limited. Malnutrition is a subacute or chronic condition related to insufficient consumption or absorption of nutrients. Malnutrition leads to changes in body composition and diminished functions, exemplified by anthropometric measures of the infant below 2 standard deviations compared to an age-matched control population. Underweight is defined by a low weight-for-age Z-score, wasted by a low weight-for-height Z-score, stunted by a low height-for-age Z-score and malnourished refers to a low mid-upper arm circumference (MUAC) for age. In a systematic review in SSA, risk factors for malnutrition were low maternal education, short birth intervals of <18 months, being first or second in birth order, male sex, lack of safe drinking water, and economic instability. On the other hand, antenatal health education could reduce the risk for malnutrition. Malnutrition is associated with detrimental infant outcomes including reduced physical growth, lower intellectual quotient, behavioral problems, and deficient social skills.

Poor water, sanitation and hygiene (WASH) affects approximately one third of the world's population. For instance, in Africa, approximately 70% of water systems are frequently non-functional and people walk long distances to collect water. On the other hand, in SSA, sewage systems are frequently inefficient with sewage bursts or lacking altogether. Lack of efficient WASH practices has been associated with intestinal infections and malnutrition in infants in SSA. The effects of WASH and malnutrition on infant development are at least partially mediated by the intestinal microbiota and the disruption of interaction networks of intestinal bacteria. From birth throughout life, human microbiome profile is constantly changing either temporarily or permanently due to diet, exposure to microbes, or medications. In birth cohorts from Bangladesh and other continents, an "ecogroup" of bacterial taxa showed consistent co-variation. Variations in this ecogroup concisely reflected microbiota development and the level of microbiota perturbation in infants with severe and moderate acute malnutrition. A causal role of the microbiota is also suggested by animal experiments. Intestinal microbiota transplantation from malnourished infants to germ-free mice resulted in a malnourished phenotype and this phenotype could even be reproduced with two isolated strains (Ruminococcus gnavus and Clostridium symbiosome). Finally, microbiota-directed complementary food corrected the intestinal microbiota of malnourished infants to a composition similar to age-matched controls, and showed superior effects in correcting growth compared to ready-to-use supplementary food.

The trajectory of the development of the intestinal microbiota is closely linked to the maturation of the infant intestinal immune system. A critical "window of opportunity" exists from birth until the end of weaning (~18 months of age), during which environmental influences can prime the immune system. In mice, a decrease in maternal epidermal growth factor intake causes the intestinal barrier to open, resulting in increased antigen passage and a vigorous immune response. This "weaning reaction" is characterized by high expression of interferon-γ (IFN-γ) and tumor necrosis factor in the intestine. Inhibition of this weaning reaction by antibiotics usage results in increased susceptibility to inflammatory conditions such as inflammatory bowel diseases (IBD) and allergies. However, how priming of the intestinal immune system is effected by environmental challenges such as infections, poor hygiene and nutrition remains unknown.

The intestinal microbiota has manifold bidirectional interactions with the host immune system. For example, Th17 cells, induced by the intestinal microbiota are a crucial line of defence against external bacteria. Further, short chain fatty acids (SCFA), and aryl hydrocarbon receptor (Ahr) agonists are microbiota products with beneficial immunomodulatory effects. Any interaction of the intestinal immune system with the microbiota should be regarded as an effort to maintain the intestinal barrier ensuring absorption of nutrients while excluding bacteria from the system and maintaining the integrity of the host.

WASH, malnutrition and associated microbiota changes lead to changes in intestinal physiology including inflammation, leakage and reduced calory absorption, which can be assessed in infants. Faecal calprotectin (FC) is an established diagnostic marker for intestinal inflammation. In the first year of life, FC values are much higher than in adulthood (277 mg/kg, vs. <50 in adults), likely related to an immature infant immune system as well as the gut microbiota. FC values decrease during the first 1.5 years of life. Variable results have been observed between 1-4 years, with possibly higher measurements in healthy infants in developing countries (Uganda).

Malnutrition has also been associated with intestinal leakage and leaky gut syndrome. Intestinal leakage leads to the loss of small and large molecules including albumin and antibodies from the systemic circulation into the gut lumen, associated with loss of calories and reduced calory absorption in the intestine. On the other hand, permeability of the intestinal wall for bacteria, bacterial toxins and/ or pathogen associated molecular patterns is increased, leading to intestinal inflammation. Intestinal leakage can be non-invasively assessed with the lactulose rhamnose permeability test.

Intestinal calory absorption can be non-invasively assessed. Bomb calorimetry can be used to measure the residual chemical energy organic material. To this end, the material will be saturated with oxygen in a sealed container and ignited, leading to the conversion of organic material to carbon dioxide, water and gaseous nitrogen. The method assesses enthalpy changes upon conversion of the organic material such as food or stool into simple gaseous molecules. Upon assessment of total energy intake with detailed food questionnaires and quantification of the residual energy in stool the total absorption capacity for energy, carbohydrates, proteins and fat has been estimated to be 89.4%, 92.5%, 86.9% and 87.3%, respectively in healthy adults.

Malnutrition is a complex condition and is also related to oral health. In African countries, inflammatory oral diseases (e.g. periodontal diseases, acute necrotising gingivitis, noma) can aggravate malnutrition due to reduced calory absorption. On the other hand, malnourishment and related conditions can also manifest as oral pathologies. Poor oral health such as missing teeth or dental caries and periodontal disease lead to diminished ability to chew or swallow certain food, leading to poorer nutritional status.

Finally, the health of the infant cannot be separated from the well-being of the mother. Mothers in low-resource settings face stress, anxiety and depression and challenges to female empowerment which might negatively impact on mother child bonding.

The current project attempts to do a comprehensive analysis of malnutrition in infants from high-density areas in Harare, Zimbabwe considering the infant microbiota, immune system, intestinal function as well as all surrounding factors affecting the health of the mother and the infant.

Rationale Gut microbiome characterization remains inadequately described in resource limited settings. In this project, investigators will recruit and follow pregnant women at high risk for subsequent malnutrition of the infant. Investigators will study development of the intestinal microbiota as well as the infant immune system, intestinal inflammation, leakage and calory extraction. This longitudinal study with comprehensive analysis of bio-samples will provide insights to move from correlation to causality. This work will inform future mechanistic studies and downstream translational work such as the development of next-generation probiotics and prebiotics.

Main hypothesis Environmental and microbiota factors result in intestinal dysfunction leading to malnutrition and suboptimal infant growth and development.

ELIGIBILITY:
Inclusion Criteria for Cases:

* MUAC ≤23 cm in pregnancy
* ≥18 years' old
* At least 20 weeks' gestational age
* Height ≥150 cm
* Planning to be staying in the study area for the next 3 years
* Willing to participate and comply with all study requirements and procedures.

Any pregnant woman meeting the above eligible criteria regardless of HIV status who meet the above inclusion criteria will be invited to participate in the study

Inclusion criteria for Controls

* Age, HIV status, gestational age at enrolment, and area residence matched normo-nourished peers with MUAC ≥25 - ≤35 cm
* Haemoglobin level of ≥11g/dL
* ≥18 years' old
* At least 20 weeks' gestational age
* Height ≥150 cm
* Planning to stay in the study area for the next 3 years

Exclusion Criteria

* Acute or chronic conditions in mothers interfering with the study according to the judgment of the investigator (HIV infection is not an exclusion criterion)
* Presence of severe mental health disorders interfering with study procedures according to the judgment of the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological
Study Population: Pregnant women at least 20 weeks gestational age seeking antenatal care services at any of the two primary health care centres, Kuwadzana and Hopely.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Alpha diversity of maternal gut microbiota | Third trimester of pregnancy, week(s) 1, 6, 14, 24, 48, 96, 144 after delivery
  Alpha diversity of maternal stool microbiota will be assessed by shotgun metagenomic sequencing, and calculated using the Shannon index. This measure reflects within-sample diversity and evenness of microbial communities.
  Unit of Measure: Shannon index (unitless; typical range 1-6)
Beta diversity of maternal gut microbiota | Third trimester of pregnancy, week(s) 1, 6, 14, 24, 48, 96, 144 after delivery
  Beta diversity of maternal stool microbiota will be assessed by shotgun metagenomic sequencing and calculated using Bray-Curtis dissimilarity. This measure reflects between-sample differences in community composition.
  Unit of Measure: % variance explained
Alpha diversity of human breast milk microbiota | Week(s) 1, 6, 14, 24, 48, 96, 144 after delivery/ until weaning
  Alpha diversity of maternal breast milk microbiota will be assessed by shotgun metagenomic sequencing, and calculated using the Shannon index. This measure reflects within-sample diversity and evenness of microbial communities.
  Unit of Measure: Shannon index (unitless; typical range 1-6)
Beta diversity of human breast milk microbiota | Week(s) 1, 6, 14, 24, 48, 96, 144 after delivery/ until weaning
  Beta diversity of breast milk microbiota will be assessed by shotgun metagenomic sequencing, and calculated using Bray-Curtis dissimilarity. This measure reflects between-sample differences in community composition. Unit of Measure: % variance explained.
Protein content of breast milk | Maternal breast milk samples collected at week(s) 1, 6, 14, 24, 48 post birth.
  Breast milk samples will be analyzed by photo-spectrometric protein assays, such as the BSA assay.
  Comparison of milk of mothers of infants with and without clinical signs of malnutrition (defined by WHO growth standards: WLZ or LAZ < -2), 100 infants per group.
  Unit of Measure: g/100mL
Fat content of breast milk | Maternal breast milk samples collected at week(s) 1, 6, 14, 24, 48 post birth.
  Breast milk samples will be analyzed by creamatocrit test. Comparison of milk of mothers of infants with and without clinical signs of malnutrition (defined by WHO growth standards: WLZ or LAZ < -2), 100 infants per group.
  Unit of Measure: mL/100mL
Lactose content of breast milk | Maternal breast milk samples collected at week(s) 1, 6, 14, 24, 48 post birth.
  Breast milk samples will be analyzed by high-performance liquid chromatography (HPLC) Comparison of milk of mothers of infants with and without clinical signs of malnutrition (defined by WHO growth standards: WLZ or LAZ < -2), 100 infants per group.
  Unit of Measure: g/100mL
Micronutrient content of breast milk | Maternal breast milk samples collected at week(s) 1, 6, 14, 24, 48 post birth.
  Breast milk micronutrients (vitamins A, D, B12, folate; trace elements such as iron, zinc, selenium) assessment using ELISA, and colorimetric assays. Comparison of milk of mothers of infants with and without clinical signs of malnutrition (defined by WHO growth standards: WLZ or LAZ < -2), 100 infants per group.
  Vit A: µg/L• Vit D: ng/mL• Folate: ng/mL• Vitamin B12: pg/mL• Iron, zinc, selenium;µg/L.
Metabolic composition of breast milk Assessing whether compositional differences in maternal milk are associated with infant intestinal development potential | Maternal breast milk samples collected at week(s) 1, 6, 14, 24, 48 post birth.
  Breast milk samples will be analyzed by untargeted mass spectrometry. Comparison of milk of mothers of infants with and without clinical signs of malnutrition (defined by WHO growth standards: WLZ or LAZ < -2), 100 infants per group.
  Unit of Measure: relative counts of ionized metabolites (mass-to-charge ratio, m/z)
Impact of breast milk on infant intestinal organoid barrier function | Maternal breast milk samples collected at week(s) 1, 6, 14, 24 post birth.
  Primary infant-derived 2D intestinal epithelial organoids will be generated from patient biopsies and treated with diluted breast milk samples to assess epithelial cell proliferation, barrier maturation, and differentiation. Transepithelial electrical resistance (TEER) will be measured as a read-out of intestinal barrier. Comparison of milk of mothers of infants with and without clinical signs of malnutrition (defined by WHO growth standards: WLZ or LAZ < -2), 100 infants per group.
  Unit of Measure: TEER: ohms·cm²
Impact of breast milk on infant intestinal organoid morphology | Maternal breast milk samples collected at week(s) 1, 6, 14, 24 post birth.
  Primary infant-derived 3D intestinal epithelial organoids will be generated from patient biopsies and treated with diluted breast milk samples for several days. Microscopy will be used to determine the organoid morphology: organoid-to-spheroid ratio. Comparison of milk of mothers of infants with and without clinical signs of malnutrition (defined by WHO growth standards: WLZ or LAZ < -2), 100 infants per group.
  Organoid morphology: villus-crypt architecture scores
  Unit of Measure: qualitative/semi-quantitative
Impact of breast milk on infant intestinal organoid size | Maternal breast milk samples collected at week(s) 1, 6, 14, 24 post birth.
  Primary infant-derived 3D intestinal epithelial organoids will be generated from patient biopsies and treated with diluted breast milk samples for several days. Microscopy will be used to determine the organoid size. Comparison of milk of mothers of infants with and without clinical signs of malnutrition (defined by WHO growth standards: WLZ or LAZ < -2), 100 infants per group.
  Unit of Measure: µm
Impact of breast milk on infant intestinal organoid gene expression | Maternal breast milk samples collected at week(s) 1, 6, 14, 24 post birth.
  Primary infant-derived 2D intestinal epithelial organoids will be generated from patient biopsies and treated with diluted breast milk samples for 24 hours. RNA will be isolated and used for reverse transcription quantitative polymerase chain reaction (RT-qPCR). Comparison of milk of mothers of infants with and without clinical signs of malnutrition (defined by WHO growth standards: WLZ or LAZ < -2), 100 infants per group.
  Expression of tight junction proteins (e.g., ZO-1, occludin): relative fluorescence intensity
  Unit of Measure: relative expression of gene of interest in relation to housekeeping gene (2^(-delta CT))
  Unit of Measure: TEER: ohms·cm²
Alpha diversity of infant gut microbiota | Week(s) 1, 6, 14, 24, 48, 96, 144 of age
  Alpha diversity of infant stool microbiota will be assessed by shotgun metagenomic sequencing, and calculated using the Shannon index. This measure reflects within-sample diversity and evenness of microbial communities.
  Unit of Measure: Shannon index (unitless; typical range 1-6)
Beta diversity of infant gut microbiota | Week(s) 1, 6, 14, 24, 48, 96, 144 of age
  Beta diversity of infant stool microbiota will be assessed by shotgun metagenomic sequencing and calculated using Bray-Curtis dissimilarity. This measure reflects between-sample differences in community composition.
  Unit of Measure: % variance explained.
Relative abundance of dominant bacterial taxa and microbial metabolic pathways | Maternal stool: third trimester, birth, 6, 12, and 24 months postpartum • Breast milk: birth, 6, and 12 months postpartum • Infant stool: birth, 6, 12, and 24 months old.
  Relative abundance of dominant bacterial taxa in maternal and infant stool, including breast milk, and of microbial metabolic pathways (KEGG modules) in infant stool, will be determined using MetaPhlAn3 and HUMAnN3.
  Unit of Measure: % of total sequences assigned.
  Relative abundance (%) of dominant bacterial taxa in maternal and infant stool
  Relative abundance (%) of microbial metabolic pathways (KEGG) in infant stool.
Maternal serum immunoglobulin concentrations | From pregnancy and once every year for 3 years
  Total IgG, IgA, and IgM will be quantified in maternal serum using ELISA/Luminex assays as biomarkers of systemic and mucosal barrier function.
  Unit of Measure: mg/mL
Maternal levels of serum proteins | From pregnancy and once every year for 3 years
  Albumin, prealbumin, and total protein will be measured in maternal serum using ELISA/Luminex assays to assess intestinal barrier integrity and nutritional status.
  Unit of Measure: g/dL
Maternal levels of serum inflammatory markers | Once in pregnancy, and once every year for 3 years.
  Myeloperoxidase, neopterin, soluble CD14, soluble CD163 and C-reactive protein will be quantified using ELISA/Luminex assays in maternal serum as biomarkers of intestinal and systemic inflammation.
  Unit of measurement: µg or ng/mL
Maternal biomarkers of epithelial and microbial translocation | Once in pregnancy, and once every year for 3 years.
  Intestinal fatty-acid binding protein (I-FABP) and endotoxin core antibodies (EndoCAb) will be measured using ELISA/Luminex assays in maternal serum as biomarkers of epithelial barrier disruption and microbial translocation.
  Unit of Measure: pg/mL (I-FABP) and EU/mL (EndoCAb).
Maternal Iron and anabolism-related biomarkers | Mother from pregnancy and once every year for 3 years
  Soluble transferrin receptor (sTfR), hepcidin, and insulin-like growth factor 1 (IGF-1) will be measured in maternal serum as biomarkers of iron status and systemic growth regulation.
  Unit of Measure: ng/mL
Maternal serum biochemical indicators | Once in pregnancy, and once every year for 3 years after delivery.
  Urea, creatinine, and liver enzyme alkaline phosphatase will be measured in maternal serum to assess renal and hepatic function.
  Unit of Measure: mg/dL (urea, creatinine) and U/L (alkaline phosphatase)
Timing of infant malnutrition and oral health status | From 6 months after delivery or birth and once a year for 2 years
  The objective is to assess the relationship between the timing of malnutrition in the infant and the development of oral health issues:
  * Dental caries
  * Oral infections and other oral manifestations,
  * Enamel dysplasia) in children from 6 months to 2 years of age.
  The standardized oral health assessment tool will be used to describe the following;
  * Dmft index (decayed, missing, filled teeth) for dental caries
  * Visual examination for enamel dysplasia
  * Oral infections including other oral manifestations
  Oral thrush (fungal) Herpetic gingivostomatitis (herpes simplex virus) Tooth abscess (bacterial) Gangrenous disease noma (bacterial) Apthous stomatitis Eruption cysts around teething teeth
Correlation between Oral Health of mother and that of the child | From 6 months after delivery or birth and once a year for 2 years
  The objective is to evaluate the correlation between the oral health status of mothers and their children, including the presence of dental caries, oral infections, and periodontal disease.
  Measurement Tool: Standardized oral health assessment tools will be used to define the following
  * DMFT index (Decayed, Missing, Filled Teeth) for mothers
  * dmft index for children
  * Plaque Index (PI) and Gingival Index (GI) for both mothers and children
  Oral health issues:
  * Dental caries
  * Oral infections and other oral manifestations,
  * Enamel dysplasia) in children from 6 months to 2 years of age.
  * Plaque/Gingival index score; Total number of surfaces with plaque/gingivitisis divided by total number of observed surfaces.
Maternal socio-demographic and the development of infant malnutrition and gut dysfunction and mortality | Mothers; from pregnancy and every 6 months until 3 years after deliveryInfants; from birth and every 6 months until 3 years old
  Determine the correlation between maternal socio-demographic, including household characteristics in pregnancy at least 20 weeks gestational age assessed using a questionnaire administered by a research nurse and,
  1. adverse pregnancy outcomes (low birth weight, pre-maturity birth < 37 weeks gestational age at birth
  2. development of infant malnutrition from birth, weeks 6, 24, 24 48, 96 and 144 of age
  3. Gut dysbiosis as in objective 1 above
  Comparing infants born of women in the 4 groups, malnourished versus normo-nourished in pregnancy at least 20 weeks gestational age by poor versus relatively better WASH living conditions Definition of malnutrition outcomes to be assessed
  * MUAC for age: Malnourished defined as those below -2SD WHO reference
  * Weight-for-age: Underweight defined as those below -2SD WHO reference
  * Weight-for-height: Wasted defined as those below -2SD WHO reference
  * Height-for-age: Stunted defined as those below -2SD WHO reference
Maternal stress assessment using Cohen Perceived Stress Scale (CPSS) | In pregnancy , weeks 6 and 24 months after delivery
  The CPSS tool measures the perception of stress in individuals and how unpredictable, uncontrollable, and overloaded mothers find their lives. It consists of 10 items with mothers rating their feelings and thoughts during the last month.
  Each item is scored 0 to 4:
  0: Never
  1. Almost never
  2. Sometimes
  3. Fairly often
  4. Very often Total Score
  The total score is calculated by summing the scores of all items, yielding a range from 0 to 40:
  Low Stress:
  Scores between 0-13. Indicates low levels of perceived stress.
  Moderate Stress:
  Scores between 14-26. Suggests moderate levels of perceived stress.
  High Stress:
  Scores between 27-40. Indicates high levels of perceived stress.
  All the 300 mothers will be assessed.
Maternal stress measurement using Edinburgh Post Partum Depression Scale (EPDS) | weeks 6 and 24 weeks and 48 weeks after delivery
  EPDS screening tool will be used to identify mothers who may be experiencing postpartum depression. It consists of 10 multiple-choice questions, each focusing on the presence or absence symptoms experienced in the past week.
  Scoring Each item on the EPDS is scored from 0 to 3, with higher scores indicating more severe symptoms. The total score can range from 0 to 30.
  Categorization of Scores 0-9: Low risk of postpartum depression. Indicates minimal or no depressive symptoms.
  10-12: Moderate risk of postpartum depression. Suggests the need for further evaluation and possibly monitoring.
  13-30: High risk of postpartum depression. Indicates significant depressive symptoms and suggests the need for further assessment and intervention.
  All the 300 mothers will be assessed.
Maternal sleeping disorders as indicator of stress using Pittsburgh Sleep Quality Index (PSQI) | In pregnancy, weeks 6 and 24 months after delivery
  The PSQI has 7 components:
  * Subjective Sleep Quality: Self-rated sleep quality.
  * Sleep latency: Time taken to fall asleep.
  * Sleep Duration: Total hours of sleep per night.
  * Habitual Sleep Efficiency: Ratio of actual sleep time to time spent in bed.
  * Frequency of problems that disrupt sleep.
  * Use of sleeping medications to aid sleep.
  * Daytime Dysfunction: Impact of sleepiness or fatigue on daily activities. Scoring Each component is scored from 0 to 3, with higher scores indicating worse sleep quality.
  Total score ranges from 0 to 21. Interpretation 0-5: Good sleep quality 6-10: Moderate sleep problems 11-21: Severe sleep problems This assessment helps in identifying mothers who may require further evaluation or intervention for sleep-related issues.
  All the 300 mothers will be assessed.
Sleeping disorders assessment using Epworth Sleepiness Scale (ESS) | In pregnancy, weeks 6 and 24 months after delivery
  Maternal sleeping disorders will be screened using The ESS tool that measures daytime sleepiness and assesses mothers' propensity to fall asleep in different situations. It consists of eight scenarios where Mothers rate their likelihood of dozing off on a scale from 0 to 3.
  Each of the eight items is scored as follows:
  0: Would never doze
  1. Slight chance of dozing
  2. Moderate chance of dozing
  3. High chance of dozing
  All the eight scenarios are summed to give a total score ranging from 0 to 24.
  Interpretation 0-10: Normal daytime sleepiness 11-12: Mild excessive daytime sleepiness 13-15: Moderate excessive daytime sleepiness 16-24: Severe excessive daytime sleepiness
  This tool helps identifying mothers who may have sleep disorders or excessive daytime sleepiness that could impact their daily functioning, including caring for their babies.
  All the 300 mothers will be assessed.
Maternal assessment of life stressful events | In pregnancy, weeks 6 and 24 months after delivery
  The Life Stressful Events Questionnaire tool will be used to assess the impact of stressful life events (frequencies and severity) on the mothers.
  Categories of stressful events:
  Personal events:
  * Death of a loved one
  * Divorce or separation
  * Serious illness or injury
  * Job loss
  * Family Events:
  * Family member illness
  * Marital problems
  * Birth of a child
  * Changes in family structure
  Social Events:
  * Moving to a new location
  * Change in social status
  * Major life transitions (e.g retirement)
  Economic Events:
  * Financial difficulties
  * Significant changes in income or employment status
  Environmental Events:
  * Natural disasters
  * Major accidents
  Higher scores or frequency of reported stressful events are typically associated with increased levels of stress and potential negative health outcomes. Tool helps identify individuals who may benefit from further support or intervention based on their stress levels.
Maternal sleep quality measurements | In pregnancy, weeks 6 and 24 months after delivery
  Sleep quality will be measured as
  * Total sleep duration (time in hours from sleep onset to final waking)
  * Sleep onset latency (time in minutes from bedtime to the first 20-minute period of sleep)
  * Sleep efficiency (ratio of total sleep duration to total time spent in bed (hours)
  Classification into 3 groups by duration of sleeping;
  -Short sleep duration: Generally defined as less than 6 hours per night. Associated with increased risks for health issues, including fatigue, cognitive impairment, and mood disorders.
  -Adequate sleep duration: Defined as 7-9 hours per night. Considered optimal for good health, cognitive function, and overall well-being.
  -Long sleep duration: Defined as more than 9 hours per night.
  Should also be considered together with other factors such as sleep efficiency, sleep disturbances etc for a more comprehensive assessment.
  All the 300 mothers will be assessed.
Maternal empowerment status using SWPER tool | In pregnancy, weeks 6 and 24 months after delivery
  The empowerment status of women may influence how they care for their infants, ultimately affecting infant mortality and morbidity.
  Domains to be assessed;
  * Social independence
  * Decision making in house hold matters
  * Attitude towards violence
  A total of 14 items in the above SWPER 3 domains will be assessed.
  Standard cut points to categorize scores into low, medium, and high levels of empowerment will be used and correlated with infant health.
  All the 300 mothers will be assessed.
Women's marital satisfaction status using Kansas tool | In pregnancy, weeks 6 and 24 months after delivery
  Marital satisfaction status of women may influence how they care for their infants, ultimately affecting infant mortality and morbidity.
  The main question; 'How satisfied are you with your marriage?' Two more related questions are also asked.
  The responses to all the 3 questions are a seven-point Likert scale (1 = 'Extremely dissatisfied'; 2 = 'Very dissatisfied'; 3 = 'Somewhat dissatisfied'; 4 = 'Mixed'; 5 = 'Somewhat satisfied'; 6 = 'Very satisfied'; 7 = 'Extremely satisfied').
  Score will range from 3 to 21, with a higher score indicating greater marital satisfaction and will be correlated with infant health.
  All the 300 mothers will be assessed.
Concentrations of infant gut intestinal inflammation | Stool samples at 12, 24, and 36 months of age
  Infant stool will be quantified using ELISA or multiplex immunoassay for the following platforms:
  * Fecal calprotectin (intestinal inflammation)
  Comparison between infants born to mothers with different nutritional statuses (MUAC ≤23 cm vs. 25-35 cm) and exposed to either improved or poor WASH environments during pregnancy. These comparisons aim to characterize the biological signatures of environmental enteric dysfunction (EED), dysbiosis, and malnutrition, in the 4 groups.
  Unit of mesurement: Fecal calprotectin: µg/g stool•
Concentrations of infant intestinal permeability | Stool samples at 12, 24, and 36 months of age •
  Infant stool will be quantified using ELISA or multiplex immunoassay for the faecal α1-antitrypsin and albumin. Biomarker concentrations will be compared between infants born to mothers with different nutritional statuses (MUAC ≤23 cm vs. 25-35 cm) and exposed to either improved or poor WASH environments during pregnancy. These comparisons aim to characterize the biological signatures of environmental enteric dysfunction (EED), dysbiosis, and malnutrition, in the 4 groups.
  Unit of measurements:
  Fecal α1-antitrypsin, albumin: mg/dL or µg/g.
Infant fecal pH and fecal fat content | Stool samples at 12, 24, and 36 months of age •
  Infant stool will be assessed for biomarkers of malabsorption and digestive efficiency. The van de Kamer test and/or non extractive method of nuclear magnetic resonance or infrared spectroscopy will be used measure fat in dried stool samples. A nitrazine paper strip will be used to measure pH of the stool samples Comparison between infants born to mothers with different nutritional statuses (MUAC ≤23 cm vs. 25-35 cm) and exposed to either improved or poor WASH environments during pregnancy. These comparisons aim to characterize the biological signatures of environmental enteric dysfunction (EED), dysbiosis, and malnutrition, in the 4 groups.
  Units of measurement; Fecal pH: pH units (1-7 scale)
  Fecal fat: % of stool mass.
Infant systemic endotoxemia from gut leakage | Stool samples at 12, 24, and 36 months of age •
  Infant serum lipopolysaccharide (LPS) will be measured using ELISA or multiplex immunoassay. Biomarker concentrations will be compared between infants born to mothers with different nutritional statuses (MUAC ≤23 cm vs. 25-35 cm) and exposed to either improved or poor WASH environments during pregnancy. These comparisons aim to characterize the biological signatures of environmental enteric dysfunction (EED), dysbiosis, and malnutrition, in the 4 groups.
  Unit of measurement; Serum LPS: ng/mL
Percentages of circulating T and B lymphocyte subsets and natural killer | Infant blood samples collected at 12, 24, and 36 months of age. Expected measures/ Unit of measures: Percentage (%) of total PBMCs per cell subset (e.g., % CD4⁺ T cells, % CD56⁺ NK cells)
  PBMCs will be isolated from peripheral blood samples of infants at 6, 12, 24, and 36 months of age. Multicolor flow cytometry will be used to quantify the percentages of :
  * CD4⁺ and CD8⁺ T lymphocytes
  * Regulatory T cells (CD4⁺CD25⁺FOXP3⁺)
  * CD19⁺ B cells
  * CD56⁺ natural killer (NK) cells Comparisons will be stratified by maternal nutritional status (MUAC ≤23 cm vs. MUAC 25-35 cm) and household water, sanitation, and hygiene (WASH) exposure (better vs. poor WASH conditions).
  Arm/Group title: Children will be assigned to 4 groups defined by maternal nutritional status (MUAC ≤23 cm vs. 25-35 cm) and household WASH conditions (improved vs. poor) at the time of pregnancy.
  Overall number of participants: 300 children
Metabolic dysregulation and vaccine immune responses in infants presenting with malnutrition | weeks 48, 96 and 144 old.
  Investigators hypothesise that there is presence of metabolic dysregulation in malnourished infants further exacerbating this condition.
  Peripheral blood mononuclear cells of malnourished babies, including their matched normo-nourished counterparts will analysed using flow cytometry to characterise natural killer (NK) cells important in early life immunity and measure fatty acid uptake (BODIPY FL C16), glucose uptake and mitochondrial mass [MitoTracker Green (MTG)]. Granzyme B and perforin levels will be correlated with mean fluorescence intensity (MFI) MTG of NKG2A+/-CD56 dim and bright NK cells.
  All malnourished babies and theirs controls will be assessed, these results will be correlated with humoural standard EPI vaccine immune responses (titres).
Short and long term relationship between presence and frequency of early life diarrhea episodes and infant malnutrition, neurodevelopment and mental health | From birth and followed up to 3 years of age
  The prevalence and incidence of diarrhea, including recovery cycles will be determined in infants born of malnourished /normonourished women in pregnancy living relatively better/poor WASH conditions. Diarrhea episodes will be defined as any episode of acute diarrhoea (≥3 passages of loose stool for 24 hours as reported by the mother) occurring before the next study visit In stool samples we will assess intestinal pathogens (viruses, parasites, bacterial pathogens).
  Plating of stool samples on McConkey agars and Enterobacteria will be further characterized using standard and advanced microbiology tools including full-length sequencing if possible.
  Intestinal helminthes ova will be assessed using Kato Katz smear of 41.7mg stool and calculate the number of egg count per 1gram stool.
Intestinal leakage of severely malnourished babies | From 1 years old up until 3 years of age
  In all severely malnourished 50% of matched infants without malnutrition, a lactulose/ rhamnose permeability test will be done.
  Weight-for-length/height below -3 standard deviations from the median with bilateral pitting edema and mid-upper arm circumference (MUAC) measurement below 110 mm in children aged 12-36, according to the World Health Organization definition of severe malnourished.
  Following drinking the sweet solution the urine will be periodically collected by the Study Gastroenterologist, and samples will stored appropriately. Mass spectrometry assessments of urine will be done in Switzerland.
Intestinal calory extraction in severely malnourished babies | Weeks 48, 96 and 144 old regardless of whether or not the babies recover from malnutrition.
  In a subset of randomly chosen infants (20 with malnutrition and 20 matched infants without malnutrition), total calory extraction will be assessed longitudinally. Following consuming a specified diet, where the weight of the food will be accurately measured mothers will collect total infant stool for 24 hours on two subsequent days, using specific diapers.
  Analysis of remaining calories in infant stool samples will be done in Bern, Switzerland where a bomb calorimetry is available.
Colonisation patterns of Clostridioides difficile in Zimbabwe and Switzerland maternal-infant dyads | From birth and followed up every 6 months up until 3 years of age
  To compare the differential impact of infant intestinal Clostridioides difficile colonization in Zimbabwe and Switzerland maternal-infant dyads.
Intestinal inflammation assessment via endoscopy | Any affected babies from one year of age
  All infants with severe malnutrition and 50% randomly selected infants with moderate malnutrition will be offered endoscopy. Gastroscopy/rectosigmoidoscopy with general anesthesia will be done by the study Gastroenterologist. During endoscopy, biopsies will be acquired for histopathological assessment by the histopathologist, as well as assessment of inflammation and the intestinal microbiota.

SECONDARY OUTCOMES:
Concentrations of anti-Gal natural antibodies and memory B cell frequencies in infant blood and stool across early life | Infant blood, serum, and stool samples at 3, 6, 12, 24, and 36 months of age.• Serum anti-Gal IgG, IgA, IgM: µg/mL• Stool anti-Gal IgA, IgM: µg/g• Memory B cell frequency specific to α-gal: % of total B cells or spot-forming units (SFU) per 10⁶ PBMCs
  Anti-Gal natural antibody levels and memory B cell responses will be characterized in infant serum, stool, and peripheral blood mononuclear cells (PBMCs) over the first three years of life. Anti-Gal IgG, IgA, and IgM concentrations will be quantified using ELISA in both serum and stool. Additionally, memory B cells specific for the α-Gal epitope will be identified and quantified by B cell ELISpot and/or flow cytometry with α-gal-conjugated tetramers or labeled glycoconjugates.
  This outcome will assess the ontogeny and maturation of the anti-Gal antibody response and its relationship with microbial colonization, nutritional status, and WASH exposure. Functional immune memory will be evaluated in the context of microbial antigen exposure and early-life health outcomes.
  Arm/Group title: Children will be assigned to one of the four groups defined by maternal nutritional status (MUAC ≤23 cm vs. 25-35 cm) and household WASH conditions (improved vs. poor) at the time of pregnancy.
Serum concentrations of anti-Gal antibodies | Infant serum samples at 3, 6, 12, 24, and 36 months of age.
  Concentrations of anti-Gal IgG, IgA, and IgM will be quantified in infant serum using ELISA to characterize the ontogeny of the anti-Gal response and its relationship with microbial colonization, nutritional status, and WASH exposure. These measurements will provide insight into the systemic development of natural antibody repertoires across early life.
  Unit of Measure: µg/mL
Stool concentrations of anti-Gal antibodies | Infant serum samples at 3, 6, 12, 24, and 36 months of age.
  Concentrations of anti-Gal IgA and IgM will be quantified in infant stool using ELISA to assess mucosal anti-Gal antibody responses. These data will reveal how gut-associated natural antibodies develop in relation to early microbial colonization and nutritional status.
  Unit of Measure: µg/g
Frequency of anti-Gal-specific memory B cells | Infant PBMCs at 12, 24, and 36 months of age.
  Frequencies of memory B cells specific to the α-Gal epitope will be quantified in infant PBMCs using B cell ELISpot and/or flow cytometry with α-Gal-conjugated tetramers or labeled glycoconjugates. This measure captures the functional development of immune memory directed against microbial glycans in early life.
  Unit of Measure: % of total B cells or spot-forming units (SFU) per 10⁶ PBMCs
Correlation of neonate mortality/morbidity and the presence of group B streptococcus (GBS) | Neonates from pregnancy up to 6 weeks of age
  Maternal under-nutrition is generally associated low birth weight which at least in murine models increases the shedding of GBS faecal load. PCR on neonate stool samples using relevant primers. Comparison GBS shedding in neonates born to malnourished women in pregnancy vs those born to their normo-nourished peers Unit of measurement: Copies GBS/gram of stool
Levels of environmental toxins, agrochemicals, microplastics, antibiotics, antiretrovirals in drinking water and soils (heavy metals) | 5 years (1.5 years of recruitment plus about 3 years of follow up after birth.
  To determine the levels of environmental toxins, agrochemicals, microplastics, antibiotics, antiretrovirals in drinking water and soils (heavy metals) and mycotoxins in foods (fermented cow milk), their impact on infants' health and development
Maternal breast milk including including urinary versus fermented cow milk aflatoxin levels | From pregnancy and 24 months after delivery (post-lactation)
  Aflatoxin B1 (AFB1) and fumonisin B1 (FB1) are toxic secondary products of fungi that frequently contaminate staple crops in resource-limited settings. Urinary aflatoxin M1 (AFM1) and FB1, biomarkers of AFB1 and FB1 exposure, respectively, will be quantified in random antenatal urine via ELISA/Luminex and correlated with adverse birth outcomes and infant growth.
  AFB1and ochratoxin A will be tested in breastmilk around delivery and once a year for 2 years/ until weaning in all the 300 women, 4 groups. Unit of measurements ng/mL.
  Aflatoxin levels will also be determined in fermented cow milk sampled during the same period.

CONTACTS AND LOCATIONS:
Overall Officials: Kerina Duri, Phd, Principal Investigator — University of Zimbabwe; Exnevia Gomo, PhD, Study Director — University of Zimbabwe
Locations (1):
- University of Zimbabwe, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Data will be anonymised prior to release for data sharing. All original data will be stored locally in the Immunology Unit for at least 10 years on appropriate electronic devices with approval for data sharing between the collaborating Institutions. All databases will be password-protected and accessible to authorised personnel only. Data users will be required to acknowledge the source of data and to ensure that the regulatory requirements of the MRCZ and other ethics regulators reviewing the projects are met. The PI through the data manager will be responsible for the overall quality and integrity of the data. Published data will be made available to other researchers upon request and verification. Additional use of data beyond thus study will be guided by the original approved study protocols and the signed participant informed consent.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When available
Access Criteria: To be advised

REFERENCES:
- [Background] Agyepong IA, Sewankambo N, Binagwaho A, Coll-Seck AM, Corrah T, Ezeh A, Fekadu A, Kilonzo N, Lamptey P, Masiye F, Mayosi B, Mboup S, Muyembe JJ, Pate M, Sidibe M, Simons B, Tlou S, Gheorghe A, Legido-Quigley H, McManus J, Ng E, O'Leary M, Enoch J, Kassebaum N, Piot P. The path to longer and healthier lives for all Africans by 2030: the Lancet Commission on the future of health in sub-Saharan Africa. Lancet. 2017 Dec 23;390(10114):2803-2859. doi: 10.1016/S0140-6736(17)31509-X. Epub 2017 Sep 13. No abstract available. PMID 28917958
- [Background] Alderman H, Behrman JR, Glewwe P, Fernald L, Walker S. Evidence of Impact of Interventions on Growth and Development during Early and Middle Childhood. In: Bundy DAP, Silva ND, Horton S, Jamison DT, Patton GC, editors. Child and Adolescent Health and Development. 3rd edition. Washington (DC): The International Bank for Reconstruction and Development / The World Bank; 2017 Nov 20. Chapter 7. Available from http://www.ncbi.nlm.nih.gov/books/NBK525234/ PMID 30212122
- [Background] Perkins JM, Kim R, Krishna A, McGovern M, Aguayo VM, Subramanian SV. Understanding the association between stunting and child development in low- and middle-income countries: Next steps for research and intervention. Soc Sci Med. 2017 Nov;193:101-109. doi: 10.1016/j.socscimed.2017.09.039. Epub 2017 Sep 22. PMID 29028557
- [Background] Smith MI, Yatsunenko T, Manary MJ, Trehan I, Mkakosya R, Cheng J, Kau AL, Rich SS, Concannon P, Mychaleckyj JC, Liu J, Houpt E, Li JV, Holmes E, Nicholson J, Knights D, Ursell LK, Knight R, Gordon JI. Gut microbiomes of Malawian twin pairs discordant for kwashiorkor. Science. 2013 Feb 1;339(6119):548-54. doi: 10.1126/science.1229000. Epub 2013 Jan 30. PMID 23363771
- [Background] Kau AL, Planer JD, Liu J, Rao S, Yatsunenko T, Trehan I, Manary MJ, Liu TC, Stappenbeck TS, Maleta KM, Ashorn P, Dewey KG, Houpt ER, Hsieh CS, Gordon JI. Functional characterization of IgA-targeted bacterial taxa from undernourished Malawian children that produce diet-dependent enteropathy. Sci Transl Med. 2015 Feb 25;7(276):276ra24. doi: 10.1126/scitranslmed.aaa4877. PMID 25717097
- [Background] Gehrig JL, Venkatesh S, Chang HW, Hibberd MC, Kung VL, Cheng J, Chen RY, Subramanian S, Cowardin CA, Meier MF, O'Donnell D, Talcott M, Spears LD, Semenkovich CF, Henrissat B, Giannone RJ, Hettich RL, Ilkayeva O, Muehlbauer M, Newgard CB, Sawyer C, Head RD, Rodionov DA, Arzamasov AA, Leyn SA, Osterman AL, Hossain MI, Islam M, Choudhury N, Sarker SA, Huq S, Mahmud I, Mostafa I, Mahfuz M, Barratt MJ, Ahmed T, Gordon JI. Effects of microbiota-directed foods in gnotobiotic animals and undernourished children. Science. 2019 Jul 12;365(6449):eaau4732. doi: 10.1126/science.aau4732. PMID 31296738
- [Background] Keats EC, Das JK, Salam RA, Lassi ZS, Imdad A, Black RE, Bhutta ZA. Effective interventions to address maternal and child malnutrition: an update of the evidence. Lancet Child Adolesc Health. 2021 May;5(5):367-384. doi: 10.1016/S2352-4642(20)30274-1. Epub 2021 Mar 7. PMID 33691083
- [Background] Humphrey JH, Mbuya MNN, Ntozini R, Moulton LH, Stoltzfus RJ, Tavengwa NV, Mutasa K, Majo F, Mutasa B, Mangwadu G, Chasokela CM, Chigumira A, Chasekwa B, Smith LE, Tielsch JM, Jones AD, Manges AR, Maluccio JA, Prendergast AJ; Sanitation Hygiene Infant Nutrition Efficacy (SHINE) Trial Team. Independent and combined effects of improved water, sanitation, and hygiene, and improved complementary feeding, on child stunting and anaemia in rural Zimbabwe: a cluster-randomised trial. Lancet Glob Health. 2019 Jan;7(1):e132-e147. doi: 10.1016/S2214-109X(18)30374-7. PMID 30554749
- [Background] Simwanza NR, Kalungwe M, Karonga T, Mtambo CMM, Ekpenyong MS, Nyashanu M. Exploring the risk factors of child malnutrition in Sub-Sahara Africa: A scoping review. Nutr Health. 2023 Mar;29(1):61-69. doi: 10.1177/02601060221090699. Epub 2022 Apr 4. PMID 35369816
- [Background] Grantham-McGregor S. A review of studies of the effect of severe malnutrition on mental development. J Nutr. 1995 Aug;125(8 Suppl):2233S-2238S. doi: 10.1093/jn/125.suppl_8.2233S. PMID 7542705
- [Background] Omidakhsh N, von Ehrenstein OS. Improved Water, Sanitation and Utilization of Maternal and Child Health Services in South Asia-An Analysis of Demographic Health Surveys. Int J Environ Res Public Health. 2021 Jul 19;18(14):7667. doi: 10.3390/ijerph18147667. PMID 34300122
- [Background] Valcourt N, Javernick-Will A, Walters J, Linden K. System Approaches to Water, Sanitation, and Hygiene: A Systematic Literature Review. Int J Environ Res Public Health. 2020 Jan 21;17(3):702. doi: 10.3390/ijerph17030702. PMID 31973179
- [Background] McDade TW. Early environments and the ecology of inflammation. Proc Natl Acad Sci U S A. 2012 Oct 16;109 Suppl 2(Suppl 2):17281-8. doi: 10.1073/pnas.1202244109. Epub 2012 Oct 8. PMID 23045646
- [Background] Guerrant RL, DeBoer MD, Moore SR, Scharf RJ, Lima AA. The impoverished gut--a triple burden of diarrhoea, stunting and chronic disease. Nat Rev Gastroenterol Hepatol. 2013 Apr;10(4):220-9. doi: 10.1038/nrgastro.2012.239. Epub 2012 Dec 11. PMID 23229327
- [Background] Raman AS, Gehrig JL, Venkatesh S, Chang HW, Hibberd MC, Subramanian S, Kang G, Bessong PO, Lima AAM, Kosek MN, Petri WA Jr, Rodionov DA, Arzamasov AA, Leyn SA, Osterman AL, Huq S, Mostafa I, Islam M, Mahfuz M, Haque R, Ahmed T, Barratt MJ, Gordon JI. A sparse covarying unit that describes healthy and impaired human gut microbiota development. Science. 2019 Jul 12;365(6449):eaau4735. doi: 10.1126/science.aau4735. PMID 31296739
- [Background] Barratt MJ, Ahmed T, Gordon JI. Gut microbiome development and childhood undernutrition. Cell Host Microbe. 2022 May 11;30(5):617-626. doi: 10.1016/j.chom.2022.04.002. PMID 35550665
- [Background] Chen RY, Mostafa I, Hibberd MC, Das S, Mahfuz M, Naila NN, Islam MM, Huq S, Alam MA, Zaman MU, Raman AS, Webber D, Zhou C, Sundaresan V, Ahsan K, Meier MF, Barratt MJ, Ahmed T, Gordon JI. A Microbiota-Directed Food Intervention for Undernourished Children. N Engl J Med. 2021 Apr 22;384(16):1517-1528. doi: 10.1056/NEJMoa2023294. Epub 2021 Apr 7. PMID 33826814
- [Background] Al Nabhani Z, Eberl G. Imprinting of the immune system by the microbiota early in life. Mucosal Immunol. 2020 Mar;13(2):183-189. doi: 10.1038/s41385-020-0257-y. Epub 2020 Jan 27. PMID 31988466
- [Background] Ivanov II, Tuganbaev T, Skelly AN, Honda K. T Cell Responses to the Microbiota. Annu Rev Immunol. 2022 Apr 26;40:559-587. doi: 10.1146/annurev-immunol-101320-011829. Epub 2022 Feb 3. PMID 35113732
- [Background] Koninckx CR, Donat E, Benninga MA, Broekaert IJ, Gottrand F, Kolho KL, Lionetti P, Miele E, Orel R, Papadopoulou A, Pienar C, Schappi MG, Wilschanski M, Thapar N. The Use of Fecal Calprotectin Testing in Paediatric Disorders: A Position Paper of the European Society for Paediatric Gastroenterology and Nutrition Gastroenterology Committee. J Pediatr Gastroenterol Nutr. 2021 Apr 1;72(4):617-640. doi: 10.1097/MPG.0000000000003046. PMID 33716293
- [Background] Hestvik E, Tumwine JK, Tylleskar T, Grahnquist L, Ndeezi G, Kaddu-Mulindwa DH, Aksnes L, Olafsdottir E. Faecal calprotectin concentrations in apparently healthy children aged 0-12 years in urban Kampala, Uganda: a community-based survey. BMC Pediatr. 2011 Feb 2;11:9. doi: 10.1186/1471-2431-11-9. PMID 21284894
- [Background] Patterson GT, Osorio EY, Peniche A, Dann SM, Cordova E, Preidis GA, Suh JH, Ito I, Saldarriaga OA, Loeffelholz M, Ajami NJ, Travi BL, Melby PC. Pathologic Inflammation in Malnutrition Is Driven by Proinflammatory Intestinal Microbiota, Large Intestine Barrier Dysfunction, and Translocation of Bacterial Lipopolysaccharide. Front Immunol. 2022 May 26;13:846155. doi: 10.3389/fimmu.2022.846155. eCollection 2022. PMID 35720380
- [Background] Mulenga C, Sviben S, Chandwe K, Amadi B, Kayamba V, Fitzpatrick JAJ, Mudenda V, Kelly P. Epithelial Abnormalities in the Small Intestine of Zambian Children With Stunting. Front Med (Lausanne). 2022 Mar 16;9:849677. doi: 10.3389/fmed.2022.849677. eCollection 2022. PMID 35372420
- [Background] Faubion WA, Camilleri M, Murray JA, Kelly P, Amadi B, Kosek MN, Enders F, Larson J, Grover M, Boe G, Dyer R, Singh R. Improving the detection of environmental enteric dysfunction: a lactulose, rhamnose assay of intestinal permeability in children aged under 5 years exposed to poor sanitation and hygiene. BMJ Glob Health. 2016 Jul 4;1(1):e000066. doi: 10.1136/bmjgh-2016-000066. eCollection 2016. PMID 28588929
- [Background] Hopper Z, Desbrow B, Roberts S, Irwin C. Preparation procedures of food and beverage samples for oxygen bomb calorimetry: A scoping review and reporting checklist. J Food Drug Anal. 2023 Jun 15;31(2):232-243. doi: 10.38212/2224-6614.3461. PMID 37335168
- [Background] Wierdsma NJ, Peters JH, van Bokhorst-de van der Schueren MA, Mulder CJ, Metgod I, van Bodegraven AA. Bomb calorimetry, the gold standard for assessment of intestinal absorption capacity: normative values in healthy ambulant adults. J Hum Nutr Diet. 2014 Apr;27 Suppl 2:57-64. doi: 10.1111/jhn.12113. Epub 2013 May 6. PMID 23647171
- [Background] Enwonwu CO, Phillips RS, Ibrahim CD, Danfillo IS. Nutrition and oral health in Africa. Int Dent J. 2004 Dec;54(6 Suppl 1):344-51. doi: 10.1111/j.1875-595x.2004.tb00010.x. PMID 15631095
- [Background] Enwonwu CO, Salako N. The periodontal disease-systemic health-infectious disease axis in developing countries. Periodontol 2000. 2012 Oct;60(1):64-77. doi: 10.1111/j.1600-0757.2012.00447.x. PMID 22909107
- [Background] Nweke M, Ukwuoma M, Adiuku-Brown AC, Ugwu P, Nseka E. Characterization and stratification of the correlates of postpartum depression in sub-Saharan Africa: A systematic review with meta-analysis. Womens Health (Lond). 2022 Jan-Dec;18:17455057221118773. doi: 10.1177/17455057221118773. PMID 36039898
- [Background] Soboka M, Feyissa GT. The impact of maternal postnatal depression on infant growth in sub-Saharan African countries: a systematic review protocol. JBI Database System Rev Implement Rep. 2016 Mar;14(3):58-67. doi: 10.11124/JBISRIR-2016-2281. PMID 27532140
- [Background] Abreha SK, Zereyesus YA. Women's Empowerment and Infant and Child Health Status in Sub-Saharan Africa: A Systematic Review. Matern Child Health J. 2021 Jan;25(1):95-106. doi: 10.1007/s10995-020-03025-y. Epub 2020 Nov 23. PMID 33226578
- [Background] O'Dea GA, Youssef GJ, Hagg LJ, Francis LM, Spry EA, Rossen L, Smith I, Teague SJ, Mansour K, Booth A, Davies S, Hutchinson D, Macdonald JA. Associations between maternal psychological distress and mother-infant bonding: a systematic review and meta-analysis. Arch Womens Ment Health. 2023 Aug;26(4):441-452. doi: 10.1007/s00737-023-01332-1. Epub 2023 Jun 15. PMID 37316760